CLINICAL TRIAL: NCT00543114
Title: A Phase I Dose Escalation Study of Lenalidomide (Revlimid) in Combination With Fludarabine-Rituximab (Rituxan) for Previously Untreated CLL/SLL
Brief Title: Dose Escalation Study of Revlimid With Fludarabine-Rituximab for CLL/SLL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of efficacy and tolerability
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Jennifer R. Brown, MD, PhD, Assistant Professor of Medicine, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-097; RV-0162
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Leukemia
Keywords: CLL; SLL; Revlimid; lenalidomide
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; fludarabine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide, fludarabine and rituximab (Experimental): Lenalidomide-Dose level will depend upon time the participant enrolls on the study: Given orally once a day for 3 weeks followed by a one week rest period fludarabine- Dose level will vary depending upon when participant enters the trial: Given intravenously for 3-5 days Rituximab- Given intravenously on Day 1 of each 28 day cycle
  Interventions: Drug: Lenalidomide; Drug: Fludarabine; Drug: Rituximab

INTERVENTIONS:
Drug: Lenalidomide — Dose level will depend upon time the participant enrolls on the study: Given orally once a day for 3 weeks followed by a one week rest period
  Other Names: Revlimid
Drug: Fludarabine — Dose level will vary depending upon when participant enters the trial: Given intravenously for 3-5 days
Drug: Rituximab — Given intravenously on Day 1 of each 28 day cycle

SUMMARY:
The purpose of this study is to determine the safety of lenalidomide (revlimid) in combination with fludarabine and rituximab and to determine the highest dose of lenalidomide that can safely be given in that combination. Lenalidomide is a drug that alters the immune system and may also interfere with the the development of tiny blood vessels that help support tumor growth. Lenalidomide is approved by the FDA for the treatment of two different blood cancers called myelodysplastic syndrome and multiple myeloma. Lenalidomide has also been studied in subjects with relapsed CLL. In this research study we are adding lenalidomide to a well-established initial therapy for CLL/SLL.

DETAILED DESCRIPTION:
* Participants will be treated in groups (cohorts) of three to six subjects per cohort. The dose of lenalidomide or fludarabine will be increased from one cohort to the next. Regardless of the treatment cohort, participants will receive treatment in cycles lasting 28 days.
* For the first 3-5 days (depending on the group), participants will be treated on an outpatient basis in the infusion room at the Dana-Farber Clinic, with fludarabine and rituximab. Fludarabine is given intravenously for 3-5 days. Rituximab is given intravenously on day 1 of each 28-day cycle. Lenalidomide is given orally once per day for 3 weeks, followed by 1 week of rest.
* Participants will be monitored very closely during the study treatment. During the first 28 day period (cycle 1), a physical exam and routine blood tests will be performed weekly. All participants in a group must finish the first 28-day treatment period before we proceed with the next group. Once started on study treatment, participants will continue for six cycles (a cycle is 28 days) of combination therapy with all three drugs. During that period they will have a physical exam and routine blood tests on day 1 of each treatment cycle, and additional blood tests on day 15 of each cycle.
* When participants complete 6 cycles of combination therapy, they will proceed with two additional months of the lenalidomide alone, for 21 out of 28 days.
* Disease response will be evaluated after 2, 6, and 8 months of study treatment. The following tests and procedures will be performed: Physical exam; blood tests; CT scans to evaluate lymph nodes; skin testing; and bone marrow biopsy if all other tests show no evidence of any remaining CLL and if the baseline bone marrow biopsy was positive
* Participants will have a physical exam and lab work every 3 months as long as their disease remains in remission.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosed with B-CLL/SLL based on the standard histologic and immunophenotypic criteria described in the WHO classification
* No prior systemic therapy for CLL/SLL, including chemotherapy or antibody therapy
* Currently needs therapy based on 1996 NCI-WG criteria
* Measurable disease
* ECOG Performance Status of 0-2
* Laboratory test results within parameters outlined in protocol
* Able to take aspirin daily as prophylactic anticoagulation

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent document
* Pregnant or breast-feeding females
* Any condition, including the presence of abnormal laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
* Use of any other experimental drug or therapy within 28 days of baseline
* Known hypersensitivity to thalidomide
* Development of erythema nodosum characterized by a desquamating rash while taking thalidomide or similar drugs
* Prior use of lenalidomide
* Concurrent use of other anti-cancer agents or treatments
* Known positive for HIV
* Chronic active Hep B patients not on prophylactic lamivudine
* Diagnosis of Mantle Cell Lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of lenalidomide in combination with fludarabine-rituximab (FR) and to determine the maximum tolerated dose in subjects with previously untreated CLL/SLL. | 2 years

SECONDARY OUTCOMES:
To determine the objective response rate and progression-free survival following lenalidomide/FR in this patient population | 2 years
To determine the improvement in ORR following two months of consolidation lenalidomide after completion of combination therapy | 2 years
To assess effects on immune function as measured by cytokine levels, T and NK cell subsets, T cell activation during therapy and DTH vaccine responses. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R. Brown, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts